CLINICAL TRIAL: NCT05545371
Title: Randomized, Blind and Positive Control Design: a Phase III Clinical Trial to Evaluate the Consistency Between Batches of 5 Doses of Freeze-dried Rabies Vaccine (Vero Cell) and the Immunogenicity and Safety of 4 Doses of Vaccine (1-1-1-1)
Brief Title: Prevention of Rabies With Four Doses of Rabies Vaccine
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Changchun Zhuoyi Biological Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ZY202106001
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Rabies Human; Antibody

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4 doses (Experimental): Inoculate rabies vaccine according to 1-1-1-1 immunization procedure
  Interventions: Biological: immunization procedures
- 5 doses (Experimental): Inoculate rabies vaccine according to 1-1-1-1-1 immunization procedure
  Interventions: Biological: immunization procedures

INTERVENTIONS:
Biological: immunization procedures — The subjects were vaccinated with rabies vaccine according to different immunization procedures

SUMMARY:
To evaluate the non inferiority of the immunogenicity of the test vaccine inoculated according to the four dose immunization program over the five dose immunization program and the batches consistency of immunogenicity according to five dose immunization procedures.

DETAILED DESCRIPTION:
* In the population aged 10-60 years, evaluate the non inferiority of the immunogenicity of the test vaccine inoculated according to the four dose immunization program (0, 3, 7, 14/28 days) over the five dose immunization program (0, 3, 7, 14, 28 days)；
* To evaluate the consistency of immunogenicity between batches of freeze-dried human rabies vaccine (Vero cell) inoculated according to five dose immunization procedures (0, 3, 7, 14, 28 days).

ELIGIBILITY:
Inclusion Criteria:

* People aged 10-60；
* Body temperature on the day of enrollment<37.3℃ (axillary temperature)

Exclusion Criteria:

* Have a history of rabies vaccine immunization or use of rabies virus passive immunization agents；
* People with congenital or acquired immunodeficiency or other autoimmune diseases；
* Female urine pregnancy test is positive, or during pregnancy and lactation, or she has a birth plan during the study period;

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2100 (Estimated)
Dates: Start 2022-06-18 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Positive conversion rate of 14 days | 6 months
  - 14 days after the first dose of inoculation, the positive conversion rate of serum neutralizing antibody.
Antibody Geometric Mean Titer (GMT) of 14 days | 6 months
  - 14 days after the first dose of inoculation, the Geometric Mean Titer (GMT) of serum neutralizing antibody .
Positive conversion rate of 42 days | 6 months
  - The seroconversion rate of serum neutralizing antibody that 42 days after the first dose of inoculation.
Advertise Events (AE) incidence within 1 month | 6 months
  - The distribution of AE incidence in different time periods (including all, within 30 minutes, 0-3 days, 0-7 days, 8-30 days) after each dose of inoculation;
Serious Adverse Events (SAE) incidence within 6 months | 12 months
  - Incidence rate of SAE within 6 months from the first dose of inoculation to the full course of inoculation.

SECONDARY OUTCOMES:
Antibody test of 28 days | 6 months
  Detection of serum neutralizing antibody 28 days after the first dose of inoculation
Antibody GMT of 42 days | 6 months
  The serum neutralized antibody GMT 42 days after the first dose of inoculation;
Antibody test within 12 months | 18months
  The serum neutralizing antibody was detected in 3 timepoints within 12 months after the whole vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Li Miao, Study Director — Changchun Zhuoyi Biological Co., Ltd
Locations (1):
- Changchun Zhuoyi Biological Co., Ltd, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Yes
safety and antibody results.
Supporting Information: Study Protocol, ICF
Time Frame: before December 2024.
Access Criteria: public to all.